CLINICAL TRIAL: NCT04572425
Title: Pilot Study to Evaluate Virtual Reality for Pain Management in Advanced Heart Failure
Brief Title: Virtual Reality for Pain Management in Advanced Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-076
Record Dates: First submitted 2020-09-03; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure，Congestive; Acute Pain; Chronic Pain
MeSH Terms: conditions — Heart Failure; Acute Pain; Chronic Pain | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided imagery (Active Comparator): 10 minutes of guided imagery (using Apple iPad and headphones, subject watches 10 minute video of a guided-imagery session depicting a peaceful walk through a forest with instrumental background music and 2-dimensional imagery)
  Interventions: Other: Guided imagery
- Virtual reality (Experimental): 10 minutes of virtual reality (using study-administered Facebook Oculus Go VR headset with headphones, subject engages with VR application Forest of Serenity (Holosphere VR®, Birmingham, UK) that features a forest environment with voice narration that can be played in a seated or fixed position.
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Guided imagery — 10 minutes of guided imagery experience delivered on tablet
  Arms: Guided imagery
Other: Virtual reality — 10 minutes of virtual reality experience delivered by Facebook Oculus Go VR device
  Arms: Virtual reality

SUMMARY:
The purpose of this research project is to evaluate the impact of virtual reality therapy on mitigating heart failure pain in hospitalized patients with heart failure and compare this impact to that of 2-dimensional guided imagery distraction therapy.

DETAILED DESCRIPTION:
Through ongoing collaborative work between the MedStar Heart and Vascular Institute Advanced Heart Failure clinical team at our hospital and the MedStar Washington Hospital Center Palliative Care team, the research team identifies hospitalized patients with a primary diagnosis of heart failure (ACC/AHA stage C or D). Subjects will be considered for enrollment in this study if able to provide consent, at least 18 years old, and report moderate-severe pain (at least 4 out of 10 where pain is rated on a Likert scale between zero and 10) in the previous 24 hours. Subjects will be excluded if they already use VR for personal use, have intractable nausea/vomiting, history of motion sickness, history of seizures or epilepsy, have cranial structure abnormalities that prevent use of VR headset, are currently enrolled in a palliative care or pain management study, and/or are on contact isolation. Institutional review board approval will be sought and informed consent will be conducted before enrolling every patient.

After consenting to participate, in addition to usual pharmacologic pain management, 128 patients should be randomized with a 1:1 ratio to receive either one 10-minute VR session, or one 10-minute 2-dimensional guided-imagery session.

VR sessions will be administered using the Facebook (Facebook Inc., Menlo Park, CA) Oculus GO VR. The VR software that will be used is the Forest of Serenity (Holosphere VR®, Birmingham, UK) application. The guided-imagery session depicts a peaceful walk through a forest with instrumental background music and 2-dimensional imagery. Patients will watch the guided imagery video on a portable tablet for 10 minutes, the same duration as the VR intervention.

Subjects in both arms will continue to receive standard pharmacologic pain management.

Because of the nature of the compared interventions, subjects and researchers cannot be blinded to intervention. Our primary outcome measure will determine the impact of distraction therapy (either VR therapy or 2-dimensional guided imagery) on self-reported pain experience. Self-reported pain experience remains the standard for clinical pain research. Secondary outcomes will measure impact of each distraction therapy on general distress level, general quality of life, and satisfaction with pain management.

Following consent and randomization, subjects will complete surveys on electronic tablets to provide baseline data on pain scores, general distress, general quality of life, and satisfaction with pain management. Pain will be assessed using the Brief Pain Inventory-Short Form (BPI-SF, modified to assess symptoms in the last 24 hours) that includes a 0-10 Likert scale for self-reported pain as well as information about pain location, quality, and interference of pain on daily living. General distress will be measured using the NCCN Distress Thermometer (a Likert scale measuring from No Distress to Extreme Distress, where "distress" is defined by the patient; we will not include the tool's associated Problem List due to overlap with other survey questions and attempt to avoid survey fatigue). General quality of life will be measured using the Functional Assessment in Chronic Illness-Therapy in Palliative Care 14-item (FACIT-Pal 14) scale that measures non-pain symptoms and general well-being.

After completion of baseline surveys, subjects will be administered either VR therapy for 10 minutes or 2-dimensional guided imagery for 10 minutes. For both arms, a member of the research team will educate the patient on the technology and assure comfort with use, remaining outside the room but nearby during the actual 10 minutes.

Following the distraction therapy, subjects will be re-surveyed BPI-SF, FACIT-Pal 14, and Distress Thermometer (Aim 1). Both groups will also be surveyed regarding acceptance of and satisfaction with the distraction therapy intervention itself and its thematic content (Aim 2). Patients randomized to VR therapy will be surveyed regarding level of immersion of the VR experience. In order to evaluate any residual effects of the distraction therapy, enrollees will be re-surveyed BPI-SF, FACIT-Pal 14, Distress Thermometer, and pain management satisfaction questions on the following day.

Our study will reach 80% power to detect a difference of 1 unit in the pain score measure between the 2 groups using a two-sample t-test with equal variance at a two-sided alpha=0.05 and assuming a within-group standard deviation of 2 for each group. Sample size calculations were conducted in PASS.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized at study institution
* primary diagnosis of ACC/AHA Stage C or D heart failure
* reports pain on 0-10 Likert scale at least 4/10 or greater

Exclusion Criteria (any of the following):

* participant already uses virtual reality for personal use
* intractable nausea/vomiting
* history of motion sickness
* history of seizures or epilepsy
* have cranial structure abnormalities that prevent use of VR headset
* currently enrolled in a palliative care or pain management study
* on contact isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Self reported pain score | Immediately after assigned intervention
  Likert scale 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Quality of life score | Immediately after assigned intervention
  Functional Assessment in Chronic Illness-Therapy in Palliative Care 14-item scale (FACIT Pal 14 scale) -- subject replies to 14 questions about quality of life issues with responses in 5-point Likert scale (0 = not at all; 4 = very much), total score range 0-56
Self reported distress | Immediately after assigned intervention
  National Comprehensive Cancer Network Distress Thermometer -- subject rates distress at that point in time on Likert scale 0-10 (0 = no distress; 10 = worst distress)
Ease of intervention ("How easy was this technology for you to use?") -- this single question designed for this study | Immediately after assigned intervention
  Single best answer to this question: subjects choose between "easy," "normal," or "difficult"
Acceptability of intervention ("Would you use this intervention again?") -- this single question designed for this study | Immediately after assigned intervention
  Single best answer: subjects choose between two choices, "Yes" or "No"

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Groninger, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart D, Mete M, Groninger H. Virtual reality for pain management in patients with heart failure: Study rationale and design. Contemp Clin Trials Commun. 2019 Oct 12;16:100470. doi: 10.1016/j.conctc.2019.100470. eCollection 2019 Dec. PMID 31650079
- [Derived] Groninger H, Stewart D, Fisher JM, Tefera E, Cowgill J, Mete M. Virtual reality for pain management in advanced heart failure: A randomized controlled study. Palliat Med. 2021 Dec;35(10):2008-2016. doi: 10.1177/02692163211041273. Epub 2021 Aug 25. PMID 34431398